CLINICAL TRIAL: NCT01786681
Title: Use of Positive Pressure in Morbidly Obese Patients Undergoing Gastroplasty
Brief Title: Use of Positive Pressure in Morbidly Obese Patients Undergoing Reduction Stomach Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Metodista de Piracicaba (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Eli Maria Pazzianotto Forti, PhD, Universidade Metodista de Piracicaba
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: Leticia2011
Record Dates: First submitted 2013-01-31; First posted 2013-02-08 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Pulmonary Atelectasis; Respiratory Tract Diseases; Pathological Conditions, Signs and Symptoms
Keywords: Morbid obesity; Bariatric Surgery; Pulmonary Atelectasis; Spirometry; Continuous Positive Airway Pressure; Physical Therapy Specialty
MeSH Terms: conditions — Pulmonary Atelectasis; Respiratory Tract Diseases; Pathological Conditions, Signs and Symptoms; Obesity, Morbid

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (4):
- Positive pressure before surgery (Experimental): Subjects treated with positive pressure in the BiPAP mode (Bi-Level Positive Airway Pressure) for one hour before bariatric surgery.
  Interventions: Procedure: Positive pressure
- Positive pressure during the surgery (Experimental): Individuals treated with 10 cm H2O of PEEP (Positive End Expiratory Pressure) during the surgical procedure.
  Interventions: Procedure: Positive pressure
- Positive pressure after surgery (Experimental): Subjects treated with positive pressure in the BiPAP mode (Bi-Level Positive Airway Pressure) for one hour after bariatric surgery.
  Interventions: Procedure: Positive pressure
- Control (No Intervention): Individuals treated with conventional physiotherapy according to the routine service of physiotherapy of the hospital.

INTERVENTIONS:
Procedure: Positive pressure
  Arms: Positive pressure after surgery; Positive pressure before surgery; Positive pressure during the surgery

SUMMARY:
The aim of this study was to investigate the effects of using positive pressure in the preoperative, intraoperative and postoperative morbidly obese individuals undergoing gastroplasty.

It is believed that the application of these devices before, during or after surgery can help to improve the lungs and reduce pulmonary complications after surgery to reduce the stomach.

DETAILED DESCRIPTION:
The aim of this study was to investigate the effects of using positive pressure in the preoperative, intraoperative and postoperative morbidly obese individuals undergoing Roux-en-Y gastric bypass with regard to: lung volumes and capacities, the prevalence of atelectasis, duration of surgery and diaphragmatic mobility.

Individuals with BMI between 40 and 55 kg/m2, aged between 25 and 55 years, were submitted to Roux-en-Y type gastric bypass by laparotomy. Patients showing a normal preoperative pulmonary function test were included, but those with hemodynamic instability, a hospital stay longer than three days or the presence of postoperative complications were excluded.

The volunteers were divided into four different groups:

Gpre: subjects treated with positive pressure in the BiPAP mode (Bi-Level Positive Airway Pressure) for one hour before surgery; Gpos: individuals treated with positive airway pressure (BiPAP) for one hour after surgery; Gpeep: individuals treated with 10 cm H2O of PEEP (Positive End Expiratory Pressure) during the surgical procedure.

Gcont: individuals treated with conventional physiotherapy (CP) according to the routine service of physiotherapy of the hospital, including the techniques of pulmonary re-expansion, breathing exercises (deep breaths or fractional), the use of incentive spirometry (Respiron®), bronchial hygiene resources if necessary (Flutter® and cough active or assisted) and assisted ambulation. It should be noted that the physiotherapist was blinded to the individual's participation in the groups, and all patients received conventional physiotherapy, independent of the group in which they were included.

The respiratory evaluation (preoperative and second postoperative days) consisted of collecting the anthropometric data, a pulmonary function test and a chest radiography (inspired and expired).

ELIGIBILITY:
Inclusion Criteria:

* BMI between 40 and 55 kg/m2
* Aged between 25 and 55 years
* Submitted to Roux-en-Y type gastric bypass by laparotomy
* Normal preoperative pulmonary function test

Exclusion Criteria:

* Hemodynamic instability
* Hospital stay longer than three days
* Presence of postoperative complications

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Pulmonary function | 2 days after surgery
  Spirometry was carried out according to the guidelines of the American Thoracic Society (ATS) and European Respiratory Society (ERS) (2005). Three types of maneuver were used in order to evaluate the lung volumes and flows: Slow Vital Capacity (SVC), Forced Vital Capacity (FVC) and Maximum Voluntary Ventilation (MVV). The maneuvers were carried out until three acceptable and reproducible curves were obtained, not exceeding more than eight attempts. The values extracted from each maneuver were selected according to Pereira (2002), and the predicted values calculated using the equation proposed by Pereira et al. (1992) for Brazilians.
Prevalence of atelectasis | 2 days after surgery
  The radiological report on the inspiration radiography, issued by the hospital radiologist, was used to analyze the presence of atelectasis.
Thoracoabdominal mobility | 2 days after surgery
  The measurement of thoracoabdominal mobility was performed by using a tape scaled in centimeters. In the standing position, the measurements were made at levels axillary, xiphoid and abdominal during rest, and at maximal inspiration and maximal expiration. At each level, the measurements were performed three times. It computed the highest value of inspiration and the lowest of expiration. The absolute difference between these values was considered the thoracoabdominal mobility.
Diaphragmatic mobility | 2 days after surgery
  The chest X-ray was made using two radiographic exposures, with the patient in the standing position. The first was taken at the end of a maximal inspiration, seeking the largest inspired lung volume (Total Lung Capacity - TLC), and the second in profound exhalation without changing the position of the film or the patient, seeking the maximum emptying of the lungs (Residual Volume - RV). The diaphragmatic motion was analyzed by superimposing the two radiological films, and calculating the distance between the highest point of the diaphragm in expiration and the highest point of the dome on bilateral inspiration.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Metodista de Piracicaba (UNIMEP), Piracicaba, São Paulo, Brazil